CLINICAL TRIAL: NCT05356559
Title: Blue Whiting Protein Hydrolysates and Sarcopenia Outcomes in Free-living, Community Dwelling Older Adults (SARCO_COMM).
Brief Title: Fish Protein Supplementation and Sarcopenia Outcomes in the Community
Acronym: SARCO_COMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ulster (Other)
Collaborators: University of Limerick (Other); Bio-Marine Ingredients Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21/EM/0140
Record Dates: First submitted 2022-03-10; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Fish protein; Fish hydrolysates; Protein supplementation; Older adults; Community; Muscle strength
MeSH Terms: conditions — Sarcopenia | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Parallel randomised control trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish protein (Active Comparator)
  Interventions: Dietary Supplement: Intervention
- Control (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Intervention — 12.5g (twice daily) Blue Whiting Protein Hydrolysates daily for 8 weeks
  Arms: Fish protein
Other: Control — Isocalorific Maltodextrin Citrus Flavoured Powder for 8 weeks
  Arms: Control

SUMMARY:
Sarcopenia is a progressive and generalised skeletal muscle disorder involving the accelerated loss of muscle mass and function that is associated with increase adverse outcomes including falls, functional decline, frailty and mortality. Diet, specifically protein has been proposed to have a role in the prevention and treatment of muscle loss in the older adult population nevertheless there is paucity of research on the effect of protein supplementation on lean body mass and other clinical outcomes in older adults.

This 2-arm parallel, double-blind, randomised, controlled dietary supplement human intervention study aims to investigate the effect of consuming 12.5g (twice daily) Blue Whiting Protein Hydrolysates daily in combination with exercise for 8 weeks on whole body lean mass tissue and measures of muscle strength and functionality in free living community dwelling older adults.

Participants (N150; 75/site (Ulster & Limerick); 75/group; 50-70 years) will be stratified by age, gender and BMI and randomly allocated to consume two sachets of either the Blue Whiting Protein Hydrolysates powder daily (12.5g at breakfast and lunch (Total 25g)), (mixed with an everyday food / drink product (provided by Ulster University) or an isocalorific maltodextrin citrus flavoured powder (Control) (mixed with an everyday food / drink product).

Assessments to be undertaken pre and post intervention include; body composition including lean tissue mass measured by DXA whole body scan (Ulster site only), Bio-Electrical Impedance Analysis (BIA), hand grip strength, a 'timed get up and go' test, 6 minute walk test, gait speed test, chair stand test, blood pressure measurements, a quality of life questionnaire, a health and lifestyle questionnaire and a physical activity questionnaire. A trained phlebotomist will obtain a 40ml max blood sample from each participant pre and post intervention. Blood samples will be used to measure markers associated with sarcopenia (serum 25(OH)D, pro inflammatory cytokine profile, full lipid profiles and kidney and liver profiles). A 4-day food diary will be collected at baseline only to determine habitual protein intake. At post intervention only, bone mineral density at the spine and hip will be measured by a DXA scanner.

Comparisons will be made (ANCOVA) between the intervention group and control group over time.

ELIGIBILITY:
Inclusion Criteria:

* Free-living, apparently healthy older adults
* Able to fast from 10pm prior to the appointment
* Aged 50-70 years at recruitment
* Not regularly taking protein supplements
* Free from serious musculoskeletal injury

Exclusion Criteria:

* Adults <50 years at recruitment
* Food allergy or intolerance that would prevent consumption of fish
* Diagnosed with any form of terminal disease or past medical history of conditions or medications that may interfere with supplementation and/or study outcomes, such as diabetes, kidney, digestive, thyroidal disease
* Cognitive impairment
* Exclusively receiving enteral or parenteral nutrition
* Currently taking any protein supplement
* Undertaking resistance exercise regularly
* Planning to lose weight/go on a special diet
* Any conditions/anomalies that could potentially interfere with the DXA
* Been advised not to undertake physical activity

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lean weight | Change over 8 weeks
  Measured by Bio-Electrical Impedance Analysis

SECONDARY OUTCOMES:
Muscle strength | Change over 8 weeks
  Measured via hand grip dynamometry
Mobility | Change over 8 weeks
  Assessed through 3 meter Timed up and go Test (time to walk 3 metre)
Exercise tolerance | Change over 8 weeks
  Six minute walk test - distance travelled over 6 minutes
Blood pressure | Change over 8 weeks
  Measured by a brachial blood pressure monitor
Walking speed | Change over 8 weeks
  Assessed by the gait speed test in a 4-meter distance
Functional fitness | Change over 8 weeks
  Assessed by time taken to perform five rises with arms crossed resting hands on their shoulders from seated.
Lean weight | Change over 8 weeks
  Measured by DXA scanner (grams) (Ulster site only)

OTHER OUTCOMES:
Lipid profile | Change over 8 weeks
  Measured by Clinical Chemistry analyzer
Vitamin D status | Change over 8 weeks
  Measured by LC-MS
Inflammation | Change over 8 weeks
  Cytokine profile measured by ELISA
Kidney function | Change over 8 weeks
  Measured by Clinical Chemistry analyzer
Liver function | Change over 8 weeks
  Measured by Clinical Chemistry analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University / Physical Education and Sport Sciences,, Coleraine / Limerick, Co.Londonderry / Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No